CLINICAL TRIAL: NCT00778609
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Group, 2-arm Study to Show Superiority of the Oral Contraceptive SH T00658ID Over Microgynon on Hormone Withdrawal-associated Symptoms After 6 Cycles of Treatment
Brief Title: Effect of a New Oral Contraceptive Pill on Hormone Related Symptoms Such as Pelvic Pain and Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91550; 310787 (Other: Company Internal); 2008-003226-42 (EudraCT Number)
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Oral Contraceptive; Headache; Pelvic Pain
Keywords: Combined Oral Contraceptives; Pelvic Pain; Headache
MeSH Terms: conditions — Headache; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027)
- Arm 2 (Active Comparator)
  Interventions: Drug: Encapsulated Microgynon + Placebo

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027) — Estradiol valerate (EV) and dienogest (DNG). Sequential 4-phasic regimen. Daily oral administration of one capsule SH T00658ID for 28 days per cycle for 6 treatment cycles no pill-free interval
  Arms: Arm 1
Drug: Encapsulated Microgynon + Placebo — Day 1 to 21; 0.03 mg ethinylestradiol (EE) + 0.15 mg levonorgestrel (LNG). Day 22 to 28 placebo
  Arms: Arm 2

SUMMARY:
The aim of the present study is to investigate whether women taking a new combined oral contraceptive pill (SH T00658ID, estradiol valerate/dienogest) experience fewer hormone withdrawal-associated symptoms such as pelvic pain or headache during their monthly cycle compared to a commonly used contraceptive pill (Microgynon).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years (inclusive) at visit 1, for smokers up to 35 years (inclusive)
* Otherwise healthy female subjects requesting contraception and currently using a levonorgestrel, gestodene or desogestrel containing oral contraceptive in a 21-day regimen and suffering from at least moderate pelvic pain, headache or both defined by an average value of >/= 35 mm for the 3 highest values on a visual analogue scale during cycle days 22-28.
* Normal or clinically insignificant cervical smear not requiring further follow up (or a normal result obtained within the last 6 months before screening)
* Able to tolerate ibuprofen and willing to use only ibuprofen supplied for the study.

Exclusion Criteria:

* Women with any contraindication for oral contraceptive use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 449 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare SH T00658ID (Qlaira) to Microgynon with regard to changes in frequency and intensity of the hormone withdrawal associated symptoms headache and pelvic pain on cycle days 22-28 combined into a single endpoint | Baseline to cycle 6

SECONDARY OUTCOMES:
Rescue medication consumption | Baseline to cycle 6
Frequency and intensity of other hormone-related symptoms (bloating or swelling, breast tenderness, and nausea or vomiting) during cycle days 22 to 28 | Baseline to cycle 6
Prevalence of individual hormone-related symptoms during cycle days 1 to 21 | Baseline to cycle 6
Prevalence of individual hormone-related symptoms during hormone-free interval, i.e. cycle days 27+28 for EV/DNG capsules and cycle days 22 to 28 for the comparator | Baseline, cycle 3 and cycle 6
Change in the average of the 3 highest VAS values of the hormone withdrawal associated symptoms pelvic pain or headache during cycle days 22 to 28 from baseline to cycle 3 | Baseline to cycle 3
Bleeding pattern and cycle control | Throughout
QoL Questionnaires: Psychological General Well-Being Index (PGWBI), Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) and Clinical Global Index (CGI) | Baseline, cycle 2 and cycle 5
AEs and SAEs. Concomitant medication. Vital signs (heart rate and blood pressure). Body weight | Throughout
General physical and gynecological examination | Screening and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (56):
- Australia (11):
  - Ashfield, New South Wales
  - Blacktown, New South Wales
  - Caringbah, New South Wales
  - Sydney, New South Wales
  - Fortitude Valley, Queensland
  - Kipparing, Queensland
  - Adelaide, South Australia
  - Norwood, South Australia
  - Clayton, Victoria
  - Nedlands, Western Australia
  - Subiaco, Western Australia
- Finland (2):
  - Helsinki
  - Kuopio
- France (11):
  - Paris, Paris
  - Brignoles
  - Maison Lafitte
  - Nancy
  - Nantes
  - Olivet
  - Paris
  - Saint-Germain-en-Laye
  - Seclin
  - Tarare
  - Toulouse
- Germany (11):
  - Rheinstetten, Baden-Wurttemberg
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Hanover, Lower Saxony
  - Bochum, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
- Mexico (4):
  - Hermosillo, Sonora
  - México, State of Mexico
  - Mexico City
  - México, D.F.
- Spain (6):
  - Benidorm, Alicante
  - Petrel, Alicante
  - Barcelona, Barcelona
  - Barcelona, Catalonia
  - Madrid, Madrid
  - Gijón, Principality of Asturias
- Switzerland (4):
  - Basel, Canton of Basel-City
  - Bern, Canton of Bern
  - Zurich, Canton of Zurich
  - Bern
- Bangkok, Thailand
- United Kingdom (6):
  - Cheadle, Cheshire
  - Northwood, Middlesex
  - Weston-super-Mare, North Somerset
  - Nottingham, Nottinghamshire
  - Glasgow, Stratchclyde
  - London

REFERENCES:
- [Derived] Macias G, Merki-Feld GS, Parke S, Mellinger U, Serrani M. Effects of a combined oral contraceptive containing oestradiol valerate/dienogest on hormone withdrawal-associated symptoms: results from the multicentre, randomised, double-blind, active-controlled HARMONY II study. J Obstet Gynaecol. 2013 Aug;33(6):591-6. doi: 10.3109/01443615.2013.800851. PMID 23919857
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/